CLINICAL TRIAL: NCT01899755
Title: A Study to Evaluate the Pharmacokinetics, Safety and Tolerability, Immunogenicity, and Pharmacodynamics of GSK2800528 in Healthy Subjects.
Brief Title: A Study to Evaluate the Pharmacokinetics (PK), Safety and Tolerability, Immunogenicity, and Pharmacodynamics (PD) of GSK2800528 in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116987
Record Dates: First submitted 2013-07-11; First posted 2013-07-15 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Psoriasis
Keywords: monoclonal antibody; healthy volunteer; TNF alpha
MeSH Terms: conditions — Psoriasis | interventions — Solutions; Injections; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- GSK2800528 Arm (Experimental): Subjects will be assigned to treatments in accordance with the randomization schedule in Cohorts 1 to 3. Treatments will be randomized with placebo in a 3:1 ratio. The final randomization code will also pre-define the sentinel subjects to ensure that of the first two subjects in each cohort, one will receive GSK2800528 and the other will receive placebo.
  Interventions: Drug: GSK2800528, solution for injection
- Placebo Arm (Placebo Comparator): Subjects will be assigned to treatments in accordance with the randomization schedule in Cohorts 1 to 3. Treatments will be randomized with placebo in a 3:1 ratio. The final randomization code will also pre-define the sentinel subjects to ensure that of the first two subjects in each cohort, one will receive GSK2800528 and the other will receive placebo.
  Interventions: Drug: Placebo (0.9% w/v Sodium Chloride), solution for injection
- Adalimumab Arm (Active Comparator): In Cohort 4, all subjects will receive adalimumab 40 mg (0.8 mL solution) as subcutaneous injection
  Interventions: Drug: Adalimumab, solution for injection

INTERVENTIONS:
Drug: GSK2800528, solution for injection — Drug will be administered at 3 different dose levels by subcutaneous injection.
  Arms: GSK2800528 Arm
Drug: Placebo (0.9% w/v Sodium Chloride), solution for injection — Subcutaneous injection of. 0.8 mL solution will be administered
  Arms: Placebo Arm
Drug: Adalimumab, solution for injection — Subcutaneous injection of 0.8 mL solution will be administered (40mg)
  Arms: Adalimumab Arm

SUMMARY:
GSK2800528 is being developed as a human anti-tumor necrosis factor (TNF) alpha monoclonal antibody (mAb) for the treatment of immune-inflammatory diseases. The study will be conducted in healthy volunteers and divided into 4 cohorts. Cohorts 1 to 3 will consist of groups of 12 subjects, 9 on active treatment (GSK2800528), and 3 on placebo. Cohort 4 will consist of a group of 9 subjects, all on active treatment (adalimumab).

ELIGIBILITY:
Inclusion Criteria:

* ALT, alkaline phosphatase and bilirubin <= 1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Average bazett's corrected QT interval (QTcB) < 450 msec, or QTcB < 480 msec in subjects with Bundle Branch Block.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included at the investigator's discretion provided the finding is unlikely to introduce additional risk factors, jeopardize study integrity, or to interfere with the study procedures.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 21.7 international unit/liter (IU/L) and oestradiol <110 picomoles/liter (pmol/L) is confirmatory. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods specified in study protocol.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods specified in study protocol.
* Body weight >= 60 kg and body mass index (BMI) within the range 19 to 31 kilogram/meter2 (kg/m2) (inclusive).

Exclusion Criteria:

* A positive pre-study Quantiferon test, Hepatitis B surface antigen, or positive Hepatitis C antibody result within 3 months of screening.
* Current or chronic history of liver or kidney disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Previous treatment with adalimumab.
* Current, or history of, cancer.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 3 months, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Travel to regions of high endemic tuberculosis/infection, as judged by the investigator or medical monitor, is prohibited from the start of screening until the final follow up visit.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Current evidence or history of bacterial, viral, or fungal infection within 7 days before dosing.
* Subject has received any type of vaccination within 21 days before dosing or will require vaccination prior to the end of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-07-10 (Actual); Primary Completion 2014-04-03 (Actual); Study Completion 2014-04-03 (Actual)

PRIMARY OUTCOMES:
Apparent systemic clearance (CL/F) of GSK2800528 | Up to Day 196
Apparent systemic clearance (CL/F) of adalimumab | Up to Day 140
Adverse event (AE) and Serious Adverse event (SAE) reporting | Up to Day 196
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, is associated with liver injury and impaired liver function.
Laboratory safety assessment for clinical chemistry parameters | Up to Day 196
  Safety data for laboratory clinical chemistry parameters including albumin, creatinine, glucose, sodium, potassium, chloride, calcium, total protein, aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyl transferase (GGT), alkaline phosphatise, total and direct bilirubin, and uric acid will be assessed
Laboratory safety assessment for hematology parameters | Up to Day 196
  Safety data for laboratory hematology parameters including platelet count, red blood cell (RBC) count, absolute white blood cell (WBC) count, reticulocyte count, hemoglobin, hematocrit, mean corpuscular volume (MCV), mean corpuscular haemoglobin concentration (MCHC), mean corpuscular haemoglobin (MCH), neutrophils, lymphocytes, monocytes, eosinophils, and basophils will be assessed.
Laboratory safety assessment for urinalysis parameters | Up to Day 196
  Safety data for laboratory urinalysis parameters including specific gravity, pH, glucose, protein, blood and ketones by dipstick , and microscopic examination will be assessed
Vital signs monitoring (blood pressure, heart rate, body temperature) | Up to Day 196
  Safety data for vital signs including blood pressure, heart rate, and body temperature will be measured
Electrocardiogram (ECG) monitoring | Up to Day 196
  Supine 12-lead ECG data will be monitored

SECONDARY OUTCOMES:
Plasma concentrations of GSK2800528 and derived pharmacokinetic parameters other than CL/F | Up to Day 196
  Blood samples for PK analysis of GSK2800528 will be collected to assess plasma concentration and derived PK parameters including maximum observed plasma concentration (Cmax), time to Cmax (tmax), area under the plasma concentration time curve [AUC(0-t) and AUC(0-infinity)], and apparent terminal phase half-life (t1/2)
Plasma concentrations of adalimumab and derived pharmacokinetic parameters other than CL/F | Up to Day 140
  Blood samples for PK analysis of adalimumab will be collected to assess plasma concentration and derived PK parameters including Cmax, tmax, AUC(0-t) and AUC(0-infinity), and t1/2
Incidence, titers, and specificity of anti-GSK2800528 antibodies. | Up to Day 196
Incidence, titers, and specificity of anti-adalimumab antibodies | Up to Day 140
Neutralising activity for samples with confirmed anti-drug antibodies | Up to Day 196

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 116987 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116987?search=study&study_ids=116987#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 116987 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116987 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116987 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116987 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116987 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116987 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116987 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register